CLINICAL TRIAL: NCT02432040
Title: Atorvastatin as Adjunctive Therapy for Chronic Plaque Type Psoriasis Versus Betamethasone Valerate Alone:A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy of Atorvastatin as Adjunctive Treatment for Chronic Plaque Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philippine Dermatological Society (Network)
Responsible Party: Principal Investigator, Sharlene Chua, Dr., Philippine Dermatological Society
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDS_PGH_2013_002
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Psoriasis
Keywords: chronic plaque psoriasis; psoriasis; atorvastatin; psoriasis area and severity index; betamethasone valerate
MeSH Terms: conditions — Psoriasis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin 40 mg once a day at night Patients asked to apply Betamethasone valerate 0.1% ointment twice a day, 3 weeks on, 1 week off, at the most
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Placebo tablets But patients are still asked to apply Betamethasone valerate 0.1% ointment twice a day, 3 weeks on, 1 week off, at the most
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin is a hydroxymethylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor used to treat dyslipidemia
  Other Names: Atopitar
  Arms: Atorvastatin
Drug: Placebo — Placebo tablets, made to look like the interventional drug
  Arms: Placebo

SUMMARY:
This study aimed to assess the efficacy and safety of atorvastatin 40 mg/day as an adjunct to betamethasone valerate 0.1% ointment applied twice daily in the treatment of patients with mild to moderate chronic plaque type psoriasis, as determined by mean reduction in PASI scores. Specific objectives included the determination and comparison of the absolute number and proportion of patients who achieved PASI-50 and the mean reductions in lipid profile (total cholesterol, HDL, LDL, triglycerides) and high-sensitivity C-reactive protein (hsCRP) measured from baseline and every month thereafter up to 6 months of treatment. This study also investigated the impact of atorvastatin treatment on the patients' quality of life as well as the association of clinical response to the lipid-lowering and anti-inflammatory effects of atorvastatin.

DETAILED DESCRIPTION:
This was a single-center, parallel-group, randomized, double-blind, placebo-controlled clinical trial. The study was conducted from February 2013 to October 2013 at a dermatology out-patient clinic in a tertiary hospital in the Philippines. Twenty-eight patients aged 19-65 years old assessed to have mild to moderate chronic plaque psoriasis, with psoriasis area and severity index (PASI) scores less than 10, were enrolled into the study and randomized into two equal treatment groups. Before participating in the study, patients were required to have a washout period of psoriasis pharmacotherapy for at least 2 months for phototherapy and systemic drugs, and 2 weeks for topical therapies.

Exclusion criteria were as follows: patients with uncontrolled hypertension, endocrine or other metabolic diseases; patients with known allergy to any of the treatments; patients with active liver disease or liver enzymes (AST and ALT) thrice the upper limit; patients with any myopathy or presence of elevated creatine kinase (CK-MM) levels; patients taking any drug that might interact with statins and those already taking statins or patients with clear indications for statin treatment; patients with impaired renal function or creatinine > 2.0 mg/dL; patients with active infection or white blood cell (WBC) > 10 and pregnant or lactating females. The study was conducted in accordance with the Declaration of Helsinki and approved by the ethics committee. Informed consent was obtained from all participants at study entry.

Patients were randomly assigned into the two groups through a computer-generated randomization table with sequencing of assignments unknown to the primary investigator. The assigned interventions were placed in sequentially-numbered, opaque envelopes, which were opened by one of the secondary investigators only after the patient had agreed to participate in the study. Patients were assigned numerical codes that were indicated in their case record forms.

Fourteen patients took atorvastatin 40 mg once a day while 14 patients took a similar-looking placebo tablet once a day. The study duration was 6 months. All patients were allowed to continue the use of betamethasone valerate 0.1% ointment twice a day for the duration of the study. Dispensing of the medications was done by a secondary investigator, while clinical assessment was done by the primary investigator who was blinded to the treatment assignments.

Patients' PASI scores, lipid profiles, aspartate aminotransferase (AST), alanine aminotransferase (ALT), hsCRP levels, and dermatology life and quality index (DLQI) scores were taken at baseline. Recording of the lipid profile, and AST, ALT values was done by another secondary investigator so that the primary investigator would not be biased by the decreasing values of the lipid profile or elevations in the AST or ALT. Photo-documentation was done throughout the study. Patients were also asked to bring their medications each visit so that the primary investigator could check for compliance. PASI scores, lipid profiles, AST, and ALT levels were monitored monthly, while DLQI scores and hsCRP levels were evaluated again after 6 months of therapy. Difference in the mean changes in PASI scores, lipid profile levels, DLQI scores, and hsCRP levels between groups were compared. Difference in the proportion of patients reaching 50% reduction in PASI scores (PASI-50) after 3 months and that after 6 months of therapy were compared. Correlation between the changes in PASI scores and the changes in lipid profile levels, as well as correlation between the changes in PASI scores and the changes in hsCRP levels were computed.

The period of observation for adverse events started from the time the subject received the first dose of the study drug until his last follow-up. Adverse event monitoring was by active query and spontaneous reporting.

Intention-to-treat analysis was the primary efficacy analysis. Patients included were those who had at least one assessment beyond baseline (Month 1). The last measurement of each randomized patient was moved forward to represent the end-of-treatment measurement at 6 months. Per-protocol analysis was the secondary efficacy analysis. All data analyses were performed using a statistical software (STATA 12.0).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild to moderate psoriasis vulgaris, chronic plaque type, with PASI score not more than 10
* Adult patients ≥ 19 years old and ≤ 65 years old
* Male or female
* Able to give consent
* Able to follow-up monthly for 6 months

Exclusion Criteria:

* Patients with PASI score ≥ 10
* Systemic therapy for psoriasis within the last two months
* Phototherapy within the last four weeks
* Known allergy to any of the treatments
* Active liver disease or liver enzymes (AST and ALT) more than 3 times the upper limit of normal
* Any myopathy or presence of elevated creatine kinase (CK-MM) levels
* Intake of any drug that might affect or interact with the study drug (e.g. fibrates, niacin, macrolide antibiotics)
* Patients already taking statins or patients with clear indications for statin treatment (i.e. coronary heart disease or disease equivalents according to the Adult Treatment Panel III Guidelines)
* Impaired renal function or creatinine > 2.0 mg/dL
* Active infection or WBC > 10
* Pregnant or lactating
* Uncontrolled hypertension, endocrine or other metabolic diseases

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharlene H Chua, Medicine, Principal Investigator — University of the Philippines-Philippine General Hospital Section of Dermatology; Ma. Lorna F Frez, Medicine, Study Director — University of the Philippines-Philippine General Hospital Section of Dermatology
Locations (1):
- University of the Philippines - Philippine General Hospital Section of Dermatology, Manila, Manila, Philippines

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from February 2013 to October 2013 at a dermatology out-patient clinic in a tertiary hospital in the Philippines. Patients diagnosed with mild to moderate chronic plaque type psoriasis were screened for eligibility.
Pre-assignment Details: Patients who were not newly diagnosed with psoriasis and already on medications were allowed to be enrolled into the study as long as they have been free of any systemic anti-psoriatic therapy for at least 2 months or free from topical steroids for at least 2 weeks.
Groups:
- Atorvastatin: Atorvastatin 40 mg once a day at night Patients asked to apply Betamethasone valerate 0.1% ointment twice a day, 3 weeks on, 1 week off, at the most
  Atorvastatin: Atorvastatin is an HMG-CoA reductase inhibitor used to treat dyslipidemia
- Placebo: Placebo tablets Patients are asked to apply Betamethasone valerate 0.1% ointment twice a day, 3 weeks on, 1 week off, at the most
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 14 | 14
Completed | 6 | 8
Not Completed | 8 | 6
Not completed — Lack of Efficacy | 3 | 0
Not completed — Lost to Follow-up | 4 | 5
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.29 (11.38) | 40.71 (12.00) | 41 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 7 | 4 | 11
PASI score [Mean (Standard Deviation); unit: units on a scale] — Psoriasis Area and Severity Index involves grading psoriatic plaques based on erythema (E), infiltration (I), desquamation (D). Severity is graded from 0-4 for each criteria (0 - none, 1 - slight, 2 - moderate, 3 - severe, and 4 - very severe). The body is divided into 4 regions, head, upper extremities, trunk, and lower extremities, and for each region, the surface area involvement is graded on a 0-6 scale (0 - 0% involvement, 1 - <10%, 2 - 10-<30%, 3 - 30-<50%, 4 - 50-<70%, 5 - 70-<90%, 6 - 90-100%).The highest potential PASI score is 72, with higher PASI scores indicating worse psoriasis.
  units on a scale | 5.49 (2.78) | 5.63 (2.52) | 5.56 (2.61)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 193.02 (34.85) | 197.73 (36.52) | 195.37 (35.11)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 126.73 (45.71) | 112.27 (45.37) | 119.50 (45.29)
LDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 125.88 (29.42) | 129.49 (29.11) | 127.69 (28.78)
HDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 46.13 (12.68) | 46.56 (13.13) | 46.34 (12.67)
High-sensitivity C-reactive protein (hsCRP) [Mean (Standard Deviation); unit: nmol/L] | 63.46 (119.43) | 39.62 (44.67) | 51.54 (89.31)
DLQI score [Mean (Standard Deviation); unit: units on a scale] — Dermatology Life Quality Index (DLQI) is a 10-item self-administered questionnaire designed to evaluate the quality of life of patients with skin diseases. Items are scored on a 4-point scale, with higher scores indicating a greater impairment in the quality of life. The total score is interpreted as follows: 0-1=no effect on patient's life, 2-5=mild effect, 6-10=moderate effect, 11-20=very large effect, and 21-30=extremely large effect.
  units on a scale | 11.50 (6.04) | 9.07 (5.84) | 10.29 (5.96)

OUTCOME MEASURES:

1. Primary Outcome: Mean Gross Change in Psoriasis Area and Severity Index (PASI) Scores From Baseline to the End of 6 Months
Description: Psoriasis Area and Severity Index involves grading psoriatic plaques based on erythema (E), infiltration (I), desquamation (D). Severity is graded from 0-4 for each criteria (0 - none, 1 - slight, 2 - moderate, 3 - severe, and 4 - very severe). The body is divided into 4 regions, head, upper extremities, trunk, and lower extremities, and for each region, the surface area involvement is graded on a 0-6 scale (0 - 0% involvement, 1 - <10%, 2 - 10-<30%, 3 - 30-<50%, 4 - 50-<70%, 5 - 70-<90%, 6 - 90-100%).The highest potential PASI score is 72, with higher PASI scores indicating worse psoriasis.
Time Frame: 6 months
Population: Intention-to-treat analysis was done. Patients with a baseline score and who had at least one reading after baseline were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | -2.15 (2.17) | -1.69 (2.36)

2. Primary Outcome: Percentage of Patients Achieving PASI-50 in Each Arm at the End of 6 Months
Description: Percentage of patients in each arm who will achieve 50% reduction in PASI scores at the end of 6 months will be compared
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
percentage of participants | 27.3 | 45.5

3. Secondary Outcome: Monthly Mean Changes in PASI Scores
Description: PASI scores were measured monthly and mean changes from baseline for each month for the whole 6-month duration of the study recorded.
Time Frame: Monthly from baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  Mean change for the first month | -0.72 (0.63) | -0.71 (0.88)
  Mean change for the second month | -1.67 (1.99) | -0.69 (1.00)
  Mean change for the third month | -2.19 (2.27) | -1.16 (1.52)
  Mean change for the fourth month | -2.10 (2.20) | -1.13 (2.05)
  Mean change for the fifth month | -2.15 (2.16) | -1.43 (2.59)
  Mean change for the sixth month | -2.15 (2.17) | -1.69 (2.36)

4. Secondary Outcome: Percentage of Patients Achieving PASI-50 at the End of 3 Months
Description: PASI-50 means at least a 50% reduction from baseline PASI score
Time Frame: 3 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 11 | 11
percentage of participants | 36.4 | 18.2

5. Secondary Outcome: Mean Change in Dermatology Life Quality Index (DLQI) Scores After 6 Months
Time Frame: 6 months
Population: The number of patients analyzed were the ones who completed the study. Intention-to-treat analysis was done.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 6 | 8
units on a scale | -6.5 (5.58) | -2.13 (6.56)

6. Secondary Outcome: Mean Change in Lipid Profile Levels
Time Frame: 6 months
Population: Intention-to-treat analysis was done. Patients who completed the study were included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 6 | 8
mg/dL
  Total cholesterol | -35.39 (47.94) | -38.32 (74.72)
  Triglycerides | -17.55 (49.93) | -5.12 (39.35)
  LDL Cholesterol | -45.18 (24.28) | -13.48 (24.02)
  HDL Cholesterol | 3.15 (5.95) | -0.69 (11.00)

7. Secondary Outcome: Mean Change in hsCRP Levels
Time Frame: 6 months
Population: Intention-to-treat analysis was done. Patients who completed the study were included since they were the only ones who had another hsCRP reading after baseline.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 6 | 8
nmol/L | -7.58 (32.92) | -5.14 (28.34)

8. Secondary Outcome: Adverse Events
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 14 | 14
participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=14) | Placebo (N=14)
Elevation in liver enzymes (Hepatobiliary disorders) | 1 (2) | 0 (0)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No